#### Egg Desensitization and induction of tolerance in Children

Principal Investigator: Moshe Ben-Shoshan MD

**McGill University Health Center** 

<u>Sub-Investigators:</u> Bruce Mazer MD McGill University Health Center

**Christine McCusker MD McGill University Health Center** 

#### 1 Proposed Research Questions

- 1. What is the rate of desensitization in children allergic to egg?
- 2. What are the predictors associated with success or failure of desensitization in children?
- 3. What are the molecular mechanisms involved in desensitization?

## 2 Research Objectives and Significance

We are proposing to initiate a study assessing desensitization for egg

This study would enable us to better determine the potential benefit of
desensitization in individuals with egg allergy.

More specifically, we will address the following research objectives:

#### **Objectives**

- A. To determine the rate of desensitization to egg..
- B. To characterize predictors of successful desensitization.
- C. To characterize molecular mechanisms involved in the process of desensitization.

#### 3. Gaps and Unmet Needs in Existing Knowledge on food desensitization

## 3.i Why do we need trials on food desensitization.

Foods are reported to be primary inciting allergens for anaphylaxis and account for 33.2% to 56% of all anaphylaxis cases. (1-4) Further, food-induced anaphylaxis hospital admissions are reported to have increased, mainly in the first 2 decades of life. (5;6)

At present, the only treatment for food allergy is to avoid the allergy-causing food, while the only treatment for an allergic reaction is prompt administration of intramuscular epinephrine. (7;8) Primary anaphylaxis prevention is based on allergen desensitization through immunotherapy and until recently was not available for food allergies. Although there are a few recent research protocols exploring desensitization for foods and although these have so far been largely successful, (9;10) up to this point there are no known guidelines describing the optimal candidate for desensitization nor are there criteria for the safest and most effective dosing schedule. Further, many of these studies have a very small sample size and do not use a control group. Hence, the efficacy of these protocols is hard to interpret (11-14) and additional larger scale randomized control studies are required.

#### 3.ii Why Egg.

Cow milk allergy (CMA) and egg allergies are the most common food allergies in children and recent reports suggest that rates of resolution are considerably lower than previous estimates. (15-17) Further, both CMA and egg allergy are associated with severe anaphylaxis<sup>(18;19)</sup> and due their ubiquitous use in our diet are almost impossible to strictly avoid. (20-22) In line with these, several studies suggest that quality of life of patients with milk/egg allergy and their families is severely impaired. (23-25)

With the support of AllerGen NCE and CIHR we have initiated in 2014 the first cross Canada study to assess milk desensitization. This study now includes almost 50 patients,

and our preliminarily results reveal an almost 80% success rate. We are now proposing to initiate an egg desensitization study based on the expertises, recruitment skills and data collected in our first 2 years of milk desensitization.

We hypothesize that there will be at least 50% improvement in the ability to tolerate egg. E.g. a child that was able to tolerate only 40 mg of merengue will be able to tolerate at least 60 mg subsequent to desensitization

The trial design is an RCT aiming to demonstrate superiority of the desensitization protocol to an avoidance strategy regarding the tolerated quantity of egg. The ratio of patients to control is 1:1. Patients will be block randomized in groups of 2 according to age and sex.

Egg allergy is the most common IgE mediated food allergy in children. Approximately 30% of children suffering from moderate to severe atopic dermatitis present an associated food allergy and egg is reported to be the major food allergen triggering IgE mediated allergic reactions in those with atopic dermatitis. (26) The major allergens in egg are known as Gal d 1-5 and include Ovomucoid which is the dominant egg allergen. (Gal d 1) and is a protease inhibitor, Ovalbumin (Gal d 2) & Ovotransferrin (Gal d3) and lysozyme (Gal d4). (27) Egg allergens are altered by heat and gastric enzymes and 55%-73% of those with egg allergy will be able to ingest cooked egg. (28,29) However, ovomucoid, the main egg allergen, is not affected by heating. (30) Different egg whites (e.g., goose, duck and turkey) were all found to contain proteins cross-reacting with most of the allergens in hen's egg white. (31) Presence of egg allergy has also major implications regarding safe administration of vaccines. Several vaccines are manufactures on egg containing media including yellow fever and Q fever and may induce an allergic reaction in those that are egg allergic. (32-35) Hence, use of rapid and effective desensitization to egg may be extremely beneficial prior to travel to yellow fever endemic areas. In addition, although

it was reported that the median age for tolerance to egg is 6 years  $\pm$  6 months, <sup>(36)</sup> recent studies suggest a lower resolution rate of 68% by age 16 years. <sup>(17)</sup>

Given the importance of egg allergy, protocols aiming to induce desensitization were recently explored. (37;38) These protocols reveal encouraging results with significantly increased thresholds to food-induced allergic reactions after oral immunotherapy in 100% of those with egg allergy. (12) Recently rush (11;13) and modified rush protocols (12) were suggested for egg but again studies exploring these protocols are limited by small sample size and by lack of controls as well as absence of methodologies assessing the molecular processes underlying these successful desensitization. It is suspected that the nature of this increased threshold is transient and reflects desensitization rather than true tolerance given that avoidance of these foods was shown to increase sensitization as well as to lower the threshold of subsequent reactivity. (39;40) In conclusion, the efficacy of the immunotherapy, extent of desensitization versus tolerance, the quantity/ frequency of allergen consumption required to maintain this effect and molecular mechanisms involved in the desensitization process are currently unknown.

#### 3. iii. Do we achieve only desensitization or do we induce also tolerance.

Desensitization refers to a change in the amount of food antigen needed to cause allergic symptoms; this state is dependent on regular antigen exposure. In contrast, *tolerance* refers to long-term immunologic changes associated with the ability to ingest a food without symptoms and without ongoing therapy. Desensitization is a worthwhile therapeutic goal as it allows individuals freedom from the risk of accidental ingestion in everyday settings; achieving long-term clinical tolerance would allow safe food ingestion

without ongoing therapy by inducing lasting immunologic changes. (41) Trials so far suggest that there might be loss of tolerance within 48 h following elimination of the food from the diet. (42) However, these trials are flawed by their small sample size (3 patients). (42) Given that more recent trials suggest that as long as participants ingested the maintenance dose of at least twice a week no allergic reactions are likely to occur (13) and given the abundance of egg products in our diet, it is crucial, to explore such an approach in a large scale clinical trial.

#### 3. iv Gaps regarding the roles of mast cells in desensitization.

Given that food desensitization is a relatively rapid process, mast cell are implicated to have a key role in this process. Compared to activated cells, desensitized Mast cells were shown to have had impaired degranulation, calcium flux, secretion of arachidonic acid products. (43) However, the effect of food desensitization on mast cells was not explored so far in clinical trials.

#### 3v. Gaps regarding the role of T regulatory cells in desensitization.

Although several studies in humans report that food allergens induce specific effector T cells, there are significant controversies between studies regarding the T cell phenotype dominating that response. Some studies report a Th2 dominated response in children with food allergies whereas Th1- responses underlie oral tolerance <sup>(44)</sup>. Other studies suggest that food antigens induce a Th2 response regardless of the presence of food allergy<sup>(45)</sup>. Further, it is proposed that Treg cells may be crucial to control food related allergic reactions. A potential suppressive role of Treg in food allergies was exemplified in both animal models <sup>(46-48)</sup> and in human studies. Increased numbers of Treg cells in

peripheral blood in children who outgrew milk allergy was reported <sup>(49;50)</sup> and decreased Treg suppression was associated with egg allergy in neonates <sup>(51)</sup>. Cord blood from offspring of atopic mothers showed fewer innate induced Treg cells and impaired suppression<sup>(52)</sup>. In line with these, an association with severe food allergy was described in patients with profound dysfunction of T reg cells that characterizes IPEX syndrome (immunodysregulation polyendocrinopathy enteropathy X-linked syndrome)<sup>(53)</sup>. In contrast 1 study looking at the number of Tregs in 10 children undergoing milk desensitization reports no enhancement of CD4+CD25+Foxp3+ T(reg) levels in peripheral blood and suggests that there is unlikely a role for long-lasting systemic immunologic changes in desensitization. However, this study is limited by a small sample size and relatively short period of follow up (6 months). <sup>(54)</sup> Additionally, data now suggests that Foxp3-ve Tregs may also play a role in tolerance.

## 3.vi Gaps regarding the role of demethylation in desensitization.

The rising incidence of food allergies is occurring more rapidly than changes to the genome sequence would allow<sup>(55)</sup> and epigenetic regulation (heritable changes in gene expression that occur in the absence of alterations in DNA sequences) may in part mediate the complex gene-by-environment interactions that can lead to asthma.<sup>(56)</sup> Experimental studies provide substantial in vitro data indicating that DNA methylation of genes critical to T-helper cell differentiation may induce polarization toward or away from an allergic phenotype. Methylation of DNA and resulting changes in chromatin structure have been shown to initiate the process by which the Th cells lose their plasticity and differentiate productively toward the Th1 versus the proallergic Th2 pattern

of cytokine gene expression. (57-59) So far no studies have explored the role of DNA methylation in short term processes such as desensitization for food allergens.

#### 3.vii. Gaps in role of allergen specific salivary IgA.

We hypothesize that development of an enhanced antigen specific mucosal IgA response is associated with reduced responses to oral antigen challenge in food allergy in children. Antigens delivered to the gastrointestinal mucosa are subject to a variety of barriers before they come into contact with effector cells such as mast cells, loaded with antigen specific IgE, that may trigger an adverse allergic reaction. Since the majority of allergic effector cells within the intestinal tract are below the epithelial barrier, and IgA is in much higher concentration than IgE, we may enhance blockade against allergic reactions in previously sensitized individuals through increases in mucosal IgA, and especially through an increased IgA:IgE ratio. While this has been examined experimentally in mice, the relationship between mucosal IgA and desensitization in the clinical setting is not defined.

#### 4. Methodological Approach/Study Design

Thirty four boys and girls with between 6 to 18 years of age, diagnosed with egg allergy will be approached by our study group. Participants will be recruited from the allergy clinic at the Montreal Children's Hospital.

**Inclusion criteria:** Children 6 years and older who satisfy all the following criteria will be included:

a. A history suggestive of immediate allergy to egg. A convincing clinical history of an IgE mediated reaction to a specific food will be defined as a minimum of 2 mild signs/symptoms or 1 moderate or 1 severe sign/symptom that was likely IgE mediated

and occurred within 120 minutes after ingestion or contact (or inhalation in the case of fish and shellfish). Reactions will be considered mild if they involve pruritus, urticaria, flushing, or rhinoconjunctivitis; moderate if they involve angioedema, throat tightness, gastrointestinal complaints, or breathing difficulties (other than wheeze); and severe if they involve wheeze, cyanosis, or circulatory collapse. (64-67)

- b. The presence of at least one of the following confirmatory tests:
- (a) Positive SPT to egg or its proteins (weal diameter 3 mm larger than that of the normal saline control). The allergens used will be commercial extracts of egg (Omega Labs, Toronto, Ontario).
- (b) Detection of serum specific IgE (>0.35 kU/L) to egg or any of its proteins (ovalbumin, ovomucoid, lysozyme and conalbumin), measured by fluorescence enzyme immunoassay (Phadia, CAP System, Uppsala, Sweden).
- (c) Positive oral challenge test to egg. Oral challenges will be performed with Meringue Powder according to the recommendations of the position paper of the European Academy of Allergology and Clinical Immunology <sup>(68)</sup> and in an open manner (appendix C). When subjective symptoms will appear (oral pruritus, abdominal discomfort), the challenge tests will be blinded.

Informed consent form signed by the parents or legal guardian (appendix B).

#### **Exclusion criteria.**

- 1. Patients who are unstable from a respiratory point of view.
- 2. Patients who present with intercurrent disease at the time of starting desensitization.

- 4. Non-IgE-mediated or non-immunological adverse reactions to egg.
- 5. Malignant or immunopathological diseases and/or severe primary or secondary immune deficiencies
- 6. Patients receiving immunosuppressor therapy.
- 7. Patients receiving β-blockers (including topical formulations).
- 8. Associated diseases contraindicating the use of epinephrine: cardiovascular disease or severe hypertension.

#### Subject Recruitment and Retention

Consent will be obtained by the study coordinator
Potential participants are referred to the study team by their treating allergist. They are given information about the study and a follow-up conversation - to review the study aims and procedures - with the study coordinator is scheduled. Typically, families of the potential participants will be given a week to review the study information. Following this, if potential participants are still interested in participating, they will meet with one of the investigators to review the potential benefits and risks of participation

It has been our experience that with this highly motivated group of participnats, it has not been necessary to implement procedures to monitor compliance.

Through a process of stratified randomization (according to sex), participants will be randomly assigned to one of 2 study groups. The first group will receive active desensitization, and the second group will not receive any treatment but will be followed up (appendix B protocols).

The desensitization protocol will be performed at the Center of Innovative medicine (CIM) as is currently done for our milk and peanut desensitization study, under the direct supervision of the medical and nursing staff, and with full cardiopulmonary resuscitation measures available for the treatment of possible allergic reactions that could occur during

the procedure. Oral and intravenous doses of diphenhydramine and intramuscular epinephrine were at the bedside at all times.

## **Desensitization to egg** . (12)

Desensitization will begin with combined challenge/rush desensitization. After placement of an intravenous catheter, 20 ml blood samples will be collected, skin prick test (SPT) to egg will be performed and 5 ml of saliva will be collected. These samples will be used to establish participants' baselines for the various biological markers being examined during the study. The modified challenge will begin with a first single dose of 0.1 mg of placebo, alternating with powdered egg white in the form of Meringue powder. After the initial dose, subjects will receive approximately doubling doses every 30 minutes until the highest tolerated single dose will be determined (see Appendix B for Challenge/Rush doses). For doses of 25 mg and greater, powdered meringue will be dispensed from individual preweighed containers.. After the initial dose, subjects will receive approximately doubling doses every 30 minutes until the highest tolerated single dose was determined. All doses will be mixed with an acceptable vehicle food chosen by the subject and his or her parent. Subjects treated for reactions will be observed for 2 hours, and if there is no evidence of an allergic reaction, they will be discharged home. Self-administered epinephrine will be provided to all patients' caregivers, along with instructions and indications for administration and education about the nature of possible reactions to OIT. To ensure there were no ill effects of the daily dosing, each subject will return to the CIM on the second day for an observed administration of the starting daily dose.

All challenges and escalation doses will take place in the Center of Innovative medicine (CIM) as is currently done for our milk and peanut desensitization study. The CIM services include equipment and medications required to monitor and treat potential reactions. The CIM nurse that will assist in the desensitization protocol is a nurse that has been trained to work in an intensive care unit. The patients will not be admitted, but will remain under observation for 7 h each day, with the possibility for increasing this period if required.

SPT with the allergens listed above will be performed on all patients before starting desensitization, and the tests will be repeated at 3, 6 and 12 months. Blood tests will be also performed to measure sIgE and sIgG, T cell phenotypes (including regulatory Tcells), salivary IgA and DNA methylation before desensitization, at 3 weeks and at 3, 6 and 12 months.

Reactions during the desensitization protocol will be classified according to the categories proposed by Perry et al. (69): mild reactions are defined when symptoms are limited to the oral mucosa or the skin; severe reactions include cardiovascular or respiratory symptoms or involvement of any four systems; all other reactions will classified as moderate, although we will consider isolated abdominal discomfort as mild when it lasted for 30 min or less (appendix C protocols).

#### **Build-up phase**

Subjects will begin daily home dosing based on the highest dose tolerated during the modified rushof powdered egg white in 1 to 2 tablespoons of baby food or other acceptable vehicle food. Home doses will be provided in individual pre-weighed containers, and subjects will be instructed to ingest 1 dose daily for 2 weeks. As long as

subjects tolerate current doses, the doses will be increased every 2 weeks (see dosing schedule Appendix B) until reaching 150 mg and then increased by 50 mg at each visit until reaching maintenance (300 mg). Dose escalations will be made at visits in the research unit to ensure that subjects tolerate increases, and subjects will be observed for at least 2 hours after increases for signs of clinical reactions. Subjects will be given diaries to track their dose-related symptoms during the study

The protocol will be individualized according to each patient's tolerance to egg:

- Mild allergic reactions will be treated when necessary and the regimen will be continued when the patient becomes asymptomatic. The previously tolerated dose will be repeated before resuming the process.
- Moderate reactions will be treated and desensitization would be restarted on the following day at the previously tolerated dose.
- Severe reactions will be treated with the necessary measures and in the appropriate department, followed by an assessment of whether to interrupt desensitization or reduce the dose on the following day to 1/10 of the dose that caused the reaction. The patients' parents will be instructed verbally and in writing about the recommendations to be followed after desensitization and how to treat possible allergic reactions. They will also given a direct telephone line for consultation. Patients will be instructed not to perform physical exercise (70;71) for 2 h after eating egg and not to take non-steroidal anti-inflammatory drugs for 3 h before or after ingestion. No special recommendations will be given for viral infections. (11) Participants will be given

symptom diaries and instructed to complete it daily to keep track of their allergic symptoms during the desensitization process.

Participants who are not able to achieve desensitization (desensitization defined as being able to tolerate the 300 mg maintenance dose) by 18 months following the initiation of the desensitization process will be considered treatment failures and discontinued from the study.

## Maintenance/ Follow-up Phase

Once subjects reached the daily dose of 300 mg, they will be instructed to take this daily for the length of the study (12 months). The subjects will be also instructed to otherwise continue an egg-elimination diet for the duration of the study. Subjects and families will be asked to complete daily home diaries to document that daily doses were taken, as well as to report accidental ingestions, problems with dose administration, or related symptoms. Follow-up visits in addition to and in conjunction with the biweekly visits for dose escalation will be planned at 3, 6, 9, 12 months from the second egg challenge. Each visit will involve a medical history and physical examination. egg specific skin prick testing (SPT), a blood draw similar to that at the challenge to measure serum egg-specific IgE and IgG concentrations, T cell penotyping and DNA methylation.

## Food challenges

One month after subjects reach the 300 mg dose, they will undergo a second food challenge to determine his or her allergenic reactivity to egg protein. Subjects will continue OIT dosing through the day before the challenge. The challenge will consist of 10 doses of powdered egg white given every 10 to 20 minutes in increasing amounts up to a total of 8 g of powdered egg white (6 g of egg protein).

After their year in the control arm, , oral desensitization will be offered to the control patients

**Variables measured.** The following variables will be measured in each patient:

A. The primary study variable will be the presence of desensitization defined by the ability to tolerate egg 1 year after the start of the trial. This is a qualitative variable with three categories: total desensitization ( 300mg of egg); partial desensitization ( 30-300mg of egg); and failed desensitization (<30 mg of egg). Only patients presenting total desensitization were regarded as being successfully desensitized.

- B. Secondary variables will be:
- 1. Number and severity of adverse reactions occurring after oral exposure to egg /milk during the desensitization and follow-up phases.

- 2. Minimum dose of egg white that triggered symptoms during the desensitization protocols or challenge tests.
  - 3. Days until desensitization was achieved, excluding weekends.
  - 4. Indices of desensitization:

SPT weal size and levels of sIgE and sIgG before desensitization, during follow-up and at the end of the study.

#### 5 Mast cell activation

Mast cell activation will be assessed through a proxy measure: the basophil activation test. This test is based on the percentage of CD63-expressing basophils detected by flowcytometry. This test is done by incubating basophils from highly sensitized atopic donors or preferably after priming them with Il3 (regardless of basophil source) (72;73) with sera from patients. We will assess the expression of CD63 on basophils after addition of egg/milk antigens respectively as well as an irrelevant antigen (gliadin and tetnus toxoid) The expression of CD63 on these cells is compared to values acquired after incubation with healthy controls and the same antigens. Values above the mean of CD63+ cells + 2 SD induced will be considered as positive. (74)

#### 6. Indices of T cell tolerance:

Levels of Treg and cytokine release at base line and uring desensitization. In order to characterise molecular pathways associated with desensitization, we will draw approximately 20 ml cc of blood from each participant and check their T cell phenotype including their Treg cells and the response to egg and milk proteins. As control the

response to an irrelevant antigen (gliadin) and to tetanus toxoid will be MEDICed. We will invite participants for annual follow ups in the first 5 years after study entry. We will also offer the desensitization to the control group at the end of the study.

#### 7. Egg specific salivary IgA

At the initial visit and at all follow-up visits, participants will be asked to produce 5 ml of saliva. Our work in previous desensitization studies has demonstrated that even children as young as 6 years can produce this volume of saliva. Egg-specific salivary IgA will be determined by ELISA

#### 5. Statistical Considerations

Given that previous studies in adults have attributed at least 50% improvement in the ability to tolerate egg  $,^{(75)}$  with an  $\alpha$  of 0.05 and a power (1-  $\beta$ ) of 0.80, a sample of 17 cases and 17 controls will be recruited. Statistical analyses will be performed using paired t-tests. A P value of <0.05 will be considered significant.

Descriptive statistics of the variables including means, standard deviations and frequencies were computed for all study variables. The concentrations of egg -sIgE and sIgG, the weal size, Mast cell, salivary IgA, T cell and DNA methylation status at the different study time-points will be compared with their baseline values using the one-sample paired t-test, and to the control using a 2 sample t-test.

Multiple regression models will be used to assess factors associated with response to desensitization (i.e. baseline demographic characteristics; gender; age; baseline basophile

activation; T cell status, baseline SPT and specific IgE, salivary IgA, and DNA methylation status,).

#### 6. Ethical Considerations

In the consent form given at study enrolment, participants will be advised that they will be randomly assigned to either desensitization treatment or observation alone for one year, (appendix B). Participants will also be advised that their data will be shared only among the study members. Participants who will be at the control group will be told that they will be offered the desensitization protocol one year after study entry.

## 7. Participant Confidentiality and Record Retention

All participants will be assigned a unique study code that will be used on all study documents. The link between the participants' code and their name will be stored on a password protected computer in the MUHC's Centre for Innovative Medicine, which is a restricted access unit. All study documents will be kept in a locked filing cabinet in the Centre for Innovative Medicine. Only members of the study team, and authorized oversight bodies will be allowed access to the study documents.

Study documents will be kept at the Centre for Innovative Medicine for two years after the end of the study, then transferred to Iron Mountain for long-term storage off-site.

All study documents will be stored for 25 years

#### 8. Research Deliverables and Milestones

| Timeframe | Deliverables | Milestones |
|-----------|--------------|------------|

| 011/17 – 03/ 18 | Develop sampling frame; ethics approval; | Ready to recruit participants |
|---|---|---|
| 03/18 -07/20 | Collect data from participants | 12 weeks of data collection in |
| | | treated participants completed |
| 07/20- 12/24 | Knowledge translation activities: | Preparation of abstracts and |
| | dissemination workshops & manuscript | manuscript |
| | preparation | |

## 9. Requirement for networking across Disciplines and Sites

Our researchers have a legacy of working across disciplines, across sites, and across sectors. For this study, we have assembled a multi-institutional research team with cross-disciplinary expertise Dr Ben-Shoshan (Montreal Children's Hospital, McGill University) and Dr Mazer (Montreal Children's Hospital) and Dr Stuart Carr (f Department of Pediatrics, University of Alberta, Edmonton, Canada)bring expertise in clinical immunology to the research team. Dr. Ann Clarke (Montreal General Hospital) will bring expertise in the field of clinical allergy and together with the co-investigator, Dr. Joseph, a biostatistician, will assisted with the study design and will supervise the statistical analyses. Dr Ciriaco Piccirillo (Departments of Microbiology & Immunology and Medicine, McGill University, Montreal, Quebec) will contribute their expertise in the areas of T cell phenotyping and DNA methylation status. Epidemiologic and

biostatistician skills are essential to undertaking this program of research and are represented in the persons of Moshe Ben-Shoshan (McGill) and Mr. Duncan Lejtenyi (both Msc in Epidemiology). Mr Duncan Lejtenyi will also be responsible for the laboratory evaluation of CD63 levels. Finally, as incorporated in our protocol, we will share the results of this research with representatives of key constituencies involved in the data collection –patients with food allergies and their families, physicians and allied professionals (e.g. nurses) through scientific meetings, our website and publications in medical journals.

#### 10. Organization of Research Team

The nominated principal applicant, Dr. Moshe Ben-Shoshan, and co-principal applicants, Dr. Bruce Mazer, will oversee all aspects of the proposed research. The collaborators, Dr Stark, Dr Piccirillo will aid in the recruitment of patients and the assessment T cells and DNA methylation status respectively.

Mr Duncan Lejtenyi, who had worked with our team in numerous studies will serve as research coordinator.

#### 11. External Research Partnerships and funding

As indicated above, external research partnerships are considered essential to the activities of our research team. We will apply to receive substantial financial support from the CIHR and from AllerGen (appendix D budget). We will work closely with client organizations such as the Anaphylaxis Canada , AAIA (allergy/Asthma Information Association), and the AQAA (Association québécoise des allergies

alimentaires). These support a cyber-society of people with food allergies and will provide support for our research activities from their limited budgets, again indicating the relevance of our research efforts to their needs.

| Name of Partner | Nature of participation | Contribut | ion (CA\$) | Letter<br>yes /no |
|---|---|---|---|---|
| | | Cash | In-kind | |
| Anaphyalxis | | | 1000 | Y |
| Canada | | | | |
| AAIA | | | 1000 | Y |
| AQAA | | | 1000 | Y |
| Total value of part | | | | |

#### References

- (1) Decker WW, Campbell RL, Manivannan V, Luke A, St Sauver JL, Weaver A et al. The etiology and incidence of anaphylaxis in Rochester, Minnesota: a report from the Rochester Epidemiology Project. J Allergy Clin Immunol 2008; 122(6):1161-5.
- (2) Bohlke K, Davis RL, DeStefano F, Marcy SM, Braun MM, Thompson RS. Epidemiology of anaphylaxis among children and adolescents enrolled in a health maintenance organization. J Allergy Clin Immunol 2004; 113(3):536-42.
- (3) Sheikh A, Alves B. Hospital admissions for acute anaphylaxis: time trend study. BMJ 2000; 320(7247):1441.
- (4) Gold MS. EpiPen epidemic or good clinical practice? J Paediatr Child Health 2003; 39(5):376-7.
- (5) Liew WK, Williamson E, Tang ML. Anaphylaxis fatalities and admissions in Australia. J Allergy Clin Immunol 2009; 123(2):434-42.
- (6) Lin RY, Anderson AS, Shah SN, Nurruzzaman F. Increasing anaphylaxis hospitalizations in the first 2 decades of life: New York State, 1990 2006. Ann Allergy Asthma Immunol 2008; 101(4):387-93.

- (7) Gold MS, Sainsbury R. First aid anaphylaxis management in children who were prescribed an epinephrine autoinjector device (EpiPen). J Allergy Clin Immunol 2000; 106(1 Pt 1):171-6.
- (8) Simons FE, Roberts JR, Gu X, Simons KJ. Epinephrine absorption in children with a history of anaphylaxis. J Allergy Clin Immunol 1998; 101(1 Pt 1):33-7.
- (9) Plaut M, Sawyer RT, Fenton MJ. Summary of the 2008 National Institute of Allergy and Infectious Diseases-US Food and Drug Administration Workshop on Food Allergy Clinical Trial Design. J Allergy Clin Immunol 2009; 124(4):671-8.
- (10) Ben Shoshan M, Clarke AE. Anaphylaxis: past, present and future. Allergy 2010.
- (11) Garcia RR, Urra JM, Feo-Brito F, Galindo PA, Borja J, Gomez E et al. Oral rush desensitization to egg: efficacy and safety. Clin Exp Allergy 2011; 41(9):1289-96.
- (12) Buchanan AD, Green TD, Jones SM, Scurlock AM, Christie L, Althage KA et al. Egg oral immunotherapy in nonanaphylactic children with egg allergy. J Allergy Clin Immunol 2007; 119(1):199-205.
- (13) Itoh N, Itagaki Y, Kurihara K. Rush specific oral tolerance induction in school-age children with severe egg allergy: one year follow up. Allergol Int 2010; 59(1):43-51.
- (14) Zapatero L, Alonso E, Fuentes V, Martinez MI. Oral desensitization in children with cow's milk allergy. J Investig Allergol Clin Immunol 2008; 18(5):389-96.
- (15) Fiocchi A, Schunemann HJ, Brozek J, Restani P, Beyer K, Troncone R et al. Diagnosis and Rationale for Action Against Cow's Milk Allergy (DRACMA): a summary report. J Allergy Clin Immunol 2010; 126(6):1119-28.
- (16) Steinke M, Fiocchi A, Kirchlechner V, Ballmer-Weber B, Brockow K, Hischenhuber C et al. Perceived food allergy in children in 10 European nations. A randomised telephone survey. Int Arch Allergy Immunol 2007; 143(4):290-5.
- (17) Savage JH, Matsui EC, Skripak JM, Wood RA. The natural history of egg allergy. J Allergy Clin Immunol 2007; 120(6):1413-7.
- (18) Calvani M, Cardinale F, Martelli A, Muraro A, Pucci N, Savino F et al. Risk factors for severe pediatric food anaphylaxis in Italy. Pediatr Allergy Immunol 2011.

- (19) Silva R, Gomes E, Cunha L, Falcao H. Anaphylaxis in children: A nine years retrospective study (2001-2009). Allergol Immunopathol (Madr ) 2011.
- (20) Boyano-Martinez T, Garcia-Ara C, Pedrosa M, Diaz-Pena JM, Quirce S. Accidental allergic reactions in children allergic to cow's milk proteins. J Allergy Clin Immunol 2009; 123(4):883-8.
- (21) Maiello N, Del Giudice MM, Capristo C, Decimo F, Santaniello F, Perrone L et al. Severe allergic reaction to lactulose in a child with milk allergy. Ann Allergy Asthma Immunol 2011; 107(1):85.
- (22) Nowak-Wegrzyn A, Shapiro GG, Beyer K, Bardina L, Sampson HA. Contamination of dry powder inhalers for asthma with milk proteins containing lactose. J Allergy Clin Immunol 2004; 113(3):558-60.
- (23) Leung TF, Yung E, Wong YS, Li CY, Wong GW. Quality-of-life assessment in Chinese families with food-allergic children. Clin Exp Allergy 2009; 39(6):890-6.
- (24) Gupta RS, Springston EE, Smith B, Kim JS, Pongracic JA, Wang X et al. Food allergy knowledge, attitudes, and beliefs of parents with food-allergic children in the United States. Pediatr Allergy Immunol 2010.
- (25) Kemp AS, Allen CW, Campbell DE. Parental perceptions in egg allergy: does egg challenge make a difference? Pediatr Allergy Immunol 2009; 20(7):648-53.
- (26) Breuer K, Heratizadeh A, Wulf A, Baumann U, Constien A, Tetau D et al. Late eczematous reactions to food in children with atopic dermatitis. Clin Exp Allergy 2004; 34(5):817-24.
- (27) Heine RG, Laske N, Hill DJ. The diagnosis and management of egg allergy. Curr Allergy Asthma Rep 2006; 6(2):145-52.
- (28) Urisu A, Ando H, Morita Y, Wada E, Yasaki T, Yamada K et al. Allergenic activity of heated and ovomucoid-depleted egg white. J Allergy Clin Immunol 1997; 100(2):171-6.
- (29) Des RA, Nguyen M, Paradis L, Primeau MN, Singer S. Tolerance to cooked egg in an egg allergic population. Allergy 2006; 61(7):900-1.
- (30) Bernhisel-Broadbent J, Dintzis HM, Dintzis RZ, Sampson HA. Allergenicity and antigenicity of chicken egg ovomucoid (Gal d III) compared with ovalbumin (Gal d I) in children with egg allergy and in mice. J Allergy Clin Immunol 1994; 93(6):1047-59.
- (31) Langeland T. A clinical and immunological study of allergy to hen's egg white. VI. Occurrence of proteins cross-reacting with allergens in hen's

- egg white as studied in egg white from turkey, duck, goose, seagull, and in hen egg yolk, and hen and chicken sera and flesh. Allergy 1983; 38(6):399-412.
- (32) Tey D, Heine RG. Egg allergy in childhood: an update. Curr Opin Allergy Clin Immunol 2009; 9(3):244-50.
- (33) Schuler JE, King WJ, Dayneka NL, Rastelli L, Marquis E, Chad Z et al. Administration of the adjuvanted pH1N1 vaccine in egg-allergic children at high risk for influenza A/H1N1 disease. Can J Public Health 2011; 102(3):196-9.
- (34) RUBIN SS. An allergic reaction following typhus-fever vaccine and yellow-fever vaccine due to egg yolk sensitivity. J Allergy 1946; 17:21-3.
- (35) Munoz-Cano R, Sanchez-Lopez J, Bartra J, Valero A. Yellow fever vaccine and egg allergy: really a problem? Allergy 2010; 65(4):533-4.
- (36) Cantani A, Micera M. Natural history of cow's milk allergy. An eight-year follow-up study in 115 atopic children. Eur Rev Med Pharmacol Sci 2004; 8(4):153-64.
- (37) Ibanez MD, Escudero C, Sanchez-Garcia S, Rodriguez del RP. Comprehensive Review of Current Knowledge on Egg Oral Immunotherapy. J Investig Allergol Clin Immunol 2015; 25(5):316-28.
- (38) Escudero C, Rodriguez del RP, Sanchez-Garcia S, Perez-Rangel I, Perez-Farinos N, Garcia-Fernandez C et al. Early sustained unresponsiveness after short-course egg oral immunotherapy: a randomized controlled study in egg-allergic children. Clin Exp Allergy 2015; 45(12):1833-43.
- (39) Jones SM, Pons L, Roberts JL, Scurlock AM, Perry TT, Kulis M et al. Clinical efficacy and immune regulation with peanut oral immunotherapy. J Allergy Clin Immunol 2009; 124(2):292-300, 300.
- (40) Morisset M, Moneret-Vautrin DA, Guenard L, Cuny JM, Frentz P, Hatahet R et al. Oral desensitization in children with milk and egg allergies obtains recovery in a significant proportion of cases. A randomized study in 60 children with cow's milk allergy and 90 children with egg allergy. Eur Ann Allergy Clin Immunol 2007; 39(1):12-9.
- (41) Varshney P, Jones SM, Scurlock AM, Perry TT, Kemper A, Steele P et al. A randomized controlled study of peanut oral immunotherapy: clinical desensitization and modulation of the allergic response. J Allergy Clin Immunol 2011; 127(3):654-60.
- (42) Rolinck-Werninghaus C, Staden U, Mehl A, Hamelmann E, Beyer K, Niggemann B. Specific oral tolerance induction with food in children: transient or persistent effect on food allergy? Allergy 2005; 60(10):1320-2.

- (43) Sancho-Serra MC, Simarro M, Castells M. Rapid IgE desensitization is antigen specific and impairs early and late mast cell responses targeting FcepsilonRI internalization. Eur J Immunol 2011; 41(4):1004-13.
- (44) Turcanu V, Maleki SJ, Lack G. Characterization of lymphocyte responses to peanuts in normal children, peanut-allergic children, and allergic children who acquired tolerance to peanuts. J Clin Invest 2003; 111(7):1065-72.
- (45) Thottingal TB, Stefura BP, Simons FE, Bannon GA, Burks W, HayGlass KT. Human subjects without peanut allergy demonstrate T cell-dependent, TH2-biased, peanut-specific cytokine and chemokine responses independent of TH1 expression. J Allergy Clin Immunol 2006; 118(4):905-14.
- (46) Takayama N, Igarashi O, Kweon MN, Kiyono H. Regulatory role of Peyer's patches for the inhibition of OVA-induced allergic diarrhea. Clin Immunol 2007; 123(2):199-208.
- (47) van Wijk F, Wehrens EJ, Nierkens S, Boon L, Kasran A, Pieters R et al. CD4+CD25+ T cells regulate the intensity of hypersensitivity responses to peanut, but are not decisive in the induction of oral sensitization. Clin Exp Allergy 2007; 37(4):572-81.
- (48) Cardoso CR, Teixeira G, Provinciatto PR, Godoi DF, Ferreira BR, Milanezi CM et al. Modulation of mucosal immunity in a murine model of foodinduced intestinal inflammation. Clin Exp Allergy 2008; 38(2):338-49.
- (49) Karlsson MR, Rugtveit J, Brandtzaeg P. Allergen-responsive CD4+CD25+ regulatory T cells in children who have outgrown cow's milk allergy. J Exp Med 2004; 199(12):1679-88.
- (50) Shreffler WG, Wanich N, Moloney M, Nowak-Wegrzyn A, Sampson HA. Association of allergen-specific regulatory T cells with the onset of clinical tolerance to milk protein. J Allergy Clin Immunol 2009; 123(1):43-52.
- (51) Smith M, Tourigny MR, Noakes P, Thornton CA, Tulic MK, Prescott SL. Children with egg allergy have evidence of reduced neonatal CD4(+)CD25(+)CD127(lo/-) regulatory T cell function. J Allergy Clin Immunol 2008; 121(6):1460-6, 1466.
- (52) Schaub B, Liu J, Hoppler S, Haug S, Sattler C, Lluis A et al. Impairment of T-regulatory cells in cord blood of atopic mothers. J Allergy Clin Immunol 2008; 121(6):1491-9, 1499.
- (53) Torgerson TR, Linane A, Moes N, Anover S, Mateo V, Rieux-Laucat F et al. Severe food allergy as a variant of IPEX syndrome caused by a deletion in a noncoding region of the FOXP3 gene. Gastroenterology 2007; 132(5):1705-17.

- (54) Mori F, Bianchi L, Pucci N, Azzari C, De MM, Novembre E. CD4+CD25+Foxp3+ T regulatory cells are not involved in oral desensitization. Int J Immunopathol Pharmacol 2010; 23(1):359-61.
- (55) Tan TH, Ellis JA, Saffery R, Allen KJ. The role of genetics and environment in the rise of childhood food allergy. Clin Exp Allergy 2011.
- (56) Miller RL, Ho SM. Environmental epigenetics and asthma: current concepts and call for studies. Am J Respir Crit Care Med 2008; 177(6):567-73.
- (57) Lee DU, Agarwal S, Rao A. Th2 lineage commitment and efficient IL-4 production involves extended demethylation of the IL-4 gene. Immunity 2002; 16(5):649-60.
- (58) Jones B, Chen J. Inhibition of IFN-gamma transcription by site-specific methylation during T helper cell development. EMBO J 2006; 25(11):2443-52.
- (59) Tykocinski LO, Hajkova P, Chang HD, Stamm T, Sozeri O, Lohning M et al. A critical control element for interleukin-4 memory expression in T helper lymphocytes. J Biol Chem 2005; 280(31):28177-85.
- (60) Camargo CA, Jr., Clark S, Kaplan MS, Lieberman P, Wood RA. Regional differences in EpiPen prescriptions in the United States: the potential role of vitamin D. J Allergy Clin Immunol 2007; 120(1):131-6.
- (61) Mullins RJ, Clark S, Camargo Jr CA. Regional variation in infant hypoallergenic formula prescriptions in Australia. Pediatr Allergy Immunol 2009.
- (62) Mullins RJ, Clark S, Camargo CA, Jr. Regional variation in epinephrine autoinjector prescriptions in Australia: more evidence for the vitamin D-anaphylaxis hypothesis. Ann Allergy Asthma Immunol 2009; 103(6):488-95.
- (63) Milner JD, Stein DM, McCarter R, Moon RY. Early infant multivitamin supplementation is associated with increased risk for food allergy and asthma. Pediatrics 2004; 114(1):27-32.
- (64) Ben-Shoshan M, Kagan RS, Alizadehfar R, Joseph L, Turnbull E, St.Pierre Yvan et al. Is the prevalence of peanut allergy increasing? A five-year follow-up study on the prevalence of peanut allergy in primary school children in Montreal. Journal of Allergy and Clinical Immunology 123[4], 783-8. 2009.

Ref Type: Journal (Full)

- (65) Hourihane JO, Kilburn SA, Dean P, Warner JO. Clinical characteristics of peanut allergy. Clin Exp Allergy 1997; 27(6):634-9.
- (66) Brown SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 2004; 114(2):371-6.

- (67) Sicherer SH, Burks AW, Sampson HA. Clinical features of acute allergic reactions to peanut and tree nuts in children. Pediatr 1998; 102(1):e6.
- (68) Bindslev-Jensen C, Ballmer-Weber BK, Bengtsson U, Blanco C, Ebner C, Hourihane J et al. Standardization of food challenges in patients with immediate reactions to foods--position paper from the European Academy of Allergology and Clinical Immunology. Allergy 2004; 59(7):690-7.
- (69) Perry TT, Matsui EC, Conover-Walker MK, Wood RA. Risk of oral food challenges. J Allergy Clin Immunol 2004; 114(5):1164-8.
- (70) Calvani M, Sopo SM. Exercise-induced anaphylaxis caused by wheat during specific oral tolerance induction. Ann Allergy Asthma Immunol 2007; 98(1):98-9.
- (71) Caminiti L, Passalacqua G, Vita D, Ruggeri P, Barberio G, Pajno GB. Food-exercise-induced anaphylaxis in a boy successfully desensitized to cow milk. Allergy 2007; 62(3):335-6.
- (72) Wedi B, Novacovic V, Koerner M, Kapp A. Chronic urticaria serum induces histamine release, leukotriene production, and basophil CD63 surface expression--inhibitory effects of anti-inflammatory drugs. J Allergy Clin Immunol 2000; 105(3):552-60.
- (73) Gentinetta T, Pecaric-Petkovic T, Wan D, Falcone FH, Dahinden CA, Pichler WJ et al. Individual IL-3 priming is crucial for consistent in vitro activation of donor basophils in patients with chronic urticaria. J Allergy Clin Immunol 2011.
- (74) Gyimesi E, Sipka S, Danko K, Kiss E, Hidvegi B, Gal M et al. Basophil CD63 expression assay on highly sensitized atopic donor leucocytes-a useful method in chronic autoimmune urticaria. Br J Dermatol 2004; 151(2):388-96.
- (75) Shertzer CL, Lookingbill DP. Effects of relaxation therapy and hypnotizability in chronic urticaria. Arch Dermatol 1987; 123(7):913-6.
- (76) Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG et al. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol 2008; 122(6):1154-60.
- (77) Caminiti L, Passalacqua G, Barberi S, Vita D, Barberio G, De Luca R et al. A new protocol for specific oral tolerance induction in children with IgE-mediated cow's milk allergy. Allergy Asthma Proc 2009; 30(4):443-8.

- (78) Martorell A, De la Hoz B, Ibanez MD, Bone J, Terrados MS, Michavila A et al. Oral desensitization as a useful treatment in 2-year-old children with cow's milk allergy. Clin Exp Allergy 2011; 41(9):1297-304.
- (79) Enrique E, Malek T, Pineda F, Palacios R, Bartra J, Tella R et al. Sublingual immunotherapy for hazelnut food allergy: a follow-up study. Ann Allergy Asthma Immunol 2008; 100(3):283-4.
- (80) Fernandez-Rivas M, Garrido FS, Nadal JA, Diaz dD, Garcia BE, Gonzalez-Mancebo E et al. Randomized double-blind, placebo-controlled trial of sublingual immunotherapy with a Pru p 3 quantified peach extract. Allergy 2009; 64(6):876-83.
- (81) Vassallo MF, Banerji A, Rudders SA, Clark S, Mullins RJ, Camargo CA, Jr. Season of birth and food allergy in children. Ann Allergy Asthma Immunol 2010; 104(4):307-13.
- (82) Pali-Scholl I, Jensen-Jarolim E. Anti-acid medication as a risk factor for food allergy. Allergy 2010.
- (83) Gourbeyre P, Denery S, Bodinier M. Probiotics, prebiotics, and synbiotics: impact on the gut immune system and allergic reactions. J Leukoc Biol 2011; 89(5):685-95.
- (84) Poole JA, Barriga K, Leung DY, Hoffman M, Eisenbarth GS, Rewers M et al. Timing of initial exposure to cereal grains and the risk of wheat allergy. Pediatrics 2006; 117(6):2175-82.
- (85) Du Toit G, Katz Y, Sasieni P, Mesher D, Maleki SJ, Fisher HR et al. Early consumption of peanuts in infancy is associated with a low prevalence of peanut allergy. J Allergy Clin Immunol 2008; 122(5):984-91.
- (86) Katz Y, Rajuan N, Goldberg MR, Eisenberg E, Heyman E, Cohen A et al. Early exposure to cow's milk protein is protective against IgE-mediated cow's milk protein allergy. J Allergy Clin Immunol 2010; 126(1):77-82.
- (87) Joseph CL, Ownby DR, Havstad SL, Woodcroft KJ, Wegienka G, Mackechnie H et al. Early complementary feeding and risk of food sensitization in a birth cohort. J Allergy Clin Immunol 2011.
- (88) Koplin JJ, Osborne NJ, Wake M, Martin PE, Gurrin LC, Robinson MN et al. Can early introduction of egg prevent egg allergy in infants? A population-based study. J Allergy Clin Immunol 2010; 126(4):807-13.
- (89) DesRoches A, Infante-Rivard C, Paradis L, Paradis J, Haddad E. Peanut allergy: is maternal transmission of antigens during pregnancy and breastfeeding a risk factor? J Investig Allergol Clin Immunol 2010; 20(4):289-94.

- (90) Sicherer SH, Wood RA, Stablein D, Lindblad R, Burks AW, Liu AH et al. Maternal consumption of peanut during pregnancy is associated with peanut sensitization in atopic infants. J Allergy Clin Immunol 2010; 126(6):1191-7.
- (91) Chung SY, Butts CL, Maleki SJ, Champagne ET. Linking peanut allergenicity to the processes of maturation, curing, and roasting. J Agric Food Chem 2003; 51(15):4273-7.
- (92) Liu GM, Cheng H, Nesbit JB, Su WJ, Cao MJ, Maleki SJ. Effects of boiling on the IgE-binding properties of tropomyosin of shrimp (Litopenaeus vannamei). J Food Sci 2010; 75(1):T1-T5.
- (93) Samson KT, Chen FH, Miura K, Odajima Y, Iikura Y, Naval RM et al. IgE binding to raw and boiled shrimp proteins in atopic and nonatopic patients with adverse reactions to shrimp. Int Arch Allergy Immunol 2004; 133(3):225-32.

## Appendix A: Disease burden and gaps.

Table 2. Primary and secondary prevention measures for food allergies<sup>a</sup>

| Trigg | Primary | Route of | Reference number | Secondary prevention | Refere |
|---|---|---|---|---|---|
| er | prevention | desensitization | | | nce |
| | | | | | number |
| Foods | Milk | PO, SL | (14;76-78) | Avoidance of allergenic food; | 154,15 |
| | Egg | PO | (11-13) | education of allergic individuals and | 5 |
| | Peanut | PO | (39) | their care-givers on importance of | |
| | Tree nut | SL | (79) | avoidance, improved labeling of | |
| | Peach | SL | (80) | prepackaged foods for allergens, | |
| | | | | wearing of Medic-Alert bracelet stating | |
| | | | | specific food allergy | |

<sup>&</sup>lt;sup>a</sup> only the most common foods, drugs and insect desensitization approaches are mentioned.

PO, Per os; SL, Sublingual; SC,

Table 2.Environmental factors associated with food allergy.

| Factor | study | Type of study | Effect | Reference |
|---|---|---|---|---|
| | | | | number |
| Season | Vassallo | Case control | Children younger than 5 years born in fall or winter had a 53% higher odds of | (81) |
| | MF | | food allergy compared with controls. | |
| Drugs | Palli- | Case control | The relative risk to develop food-specific IgE after anti-acid therapy was 10.5 | (82) |
| | Scholl | | (95% CI,1.44,76.48). | |
| Microbia | Gourbeyr | Review of case | No clear conclusion regarding probiotic beneficial effects on the prevention or | (83) |
| 1 exposure | e | control and cohort | treatment of allergy . | |
| | | studies | | |
| Food | Poole JA | Cohort | After adjusting for breastfeeding duration, introduction of rice cereal, family | (84) |
| consumption | | | history of allergy, and history of food allergy before 6 months of age, age at initial | |
| (quantity | | | exposure to cereal grains continued to be strongly associated with wheat allergy | |
| and timing) | | | (≥7 months: adjusted OR: 3.8; 95% CI, 1.18,12.28) | |

| Du Toit | Case control | After adjustment for atopy, other food allergies, age, and sex, the RR for | (85) |
|---|---|---|---|
| | | peanut allergy in the UK vs Israel is 5.8 (95% CI, 2.8,11.8), and largest and most | |
| | | significant difference in weaning between the UK and Israel was observed in the | |
| | | age of introduction of peanut (P < .0001). By 9 months of age, 69% of Israelis | |
| | | were eating peanut compared with only 10% of UK infants. | |
| Katz | Cohort | The OR was 19.3 (95% CI, 6.0,62.1) for development of IgE mediated CMA | (86) |
| | | among infants with exposure to cow milk protein at the age of 15 days or more (P | |
| | | < .001) vs those introduced to cow milk protein before 15 days. | |
| Joseph | Cohort | Early feeding reduced the risk of peanut sensitization among children with a | (87) |
| | | parental history [adjusted OR, 0.2 (95% CI, 0.1,0.7); P = .007]. The relationship | |
| | | also became significant for egg when a cutoff for IgE of ≥0.70 IU/mL was used | |
| | | [adjustedOR, 0.5 (95% CI, 0.3,0.9)]. | |
| Koplin | Case control | Introduction of cooked egg at age 4 to 6 months, vs later exposure reduced | (88) |
| | | the risk of egg allergy [OR, 0.2 (95% CI, 0.06-0.71)]. | |
| Des | Case control | The reported consumption of peanuts during pregnancy and breastfeeding was | (89) |
| Roches | | higher in the case group (those who developed peanut allergy and associated with | |
| | | an increased risk of peanut allergy in offspring [OR, 4.22 (95%CI, 1.57,11.30) | |
| | | and OR, 2.28 (95% CI, 1.31,3.97) for pregnancy and breastfeeding, respectively]. | |

| Sicherer | Case control | Multivariate analysis including clinical, laboratory, and demographic variables | (90) |
|---|---|---|---|
| 1 | | showed frequent peanut consumption during pregnancy {OR, 2.9(95% CI, | |
| 1 | | 1.7,4.9)] to be associated with peanut IgE ≥5 kUA/L. | |
| Chung | Laboratory analysis | After curing and roasting, mature peanuts exhibited approximately 20% higher | (91) |
| 1 | | levels of advanced glycation end adducts and higher IgE binding vs immature | |
| ı | | peanuts. | |
| Yadzir | Laboratory analysis | Extracts from raw shrimp bound higher IgE than extracts from boiled shrimp, | (92) |
| 1 | | but the purified boiled tropomysoin (the main shrimp allergen) demonstrates | |
| ı | | higher IgE binding vs raw shrimp. | |
| Samson | Laboratory | Thermal processing can lead to the formation of new antigenic structures. | (93) |
| 1 | analysis | | |
| Milner | Cohort | Early vitamin D use (within the first 6 months of life) was associated with a | (63) |
| ı | | higher risk for food allergies in the exclusively formula-fed population [OR,1.63( | |
| ı | | 95% CI,1.21,2.20)]. Vitamin use at 3 years of age was associated with increased | |
| ı | | risk for food allergies but not asthma in both breastfed [OR,1.62(95% | |
| ı | | CI,1.19,2.21) ]and exclusively formula-fed infants [OR, 1.39( 95% CI,1.03,1.88)]. | |
| ı | | | |
| Cramago | Ecologic study | Strong north-south gradient for the prescription of EpiPens in the United | (60) |
| | Chung Yadzir Samson Milner | Chung Laboratory analysis Yadzir Laboratory analysis Samson Laboratory analysis Milner Cohort | showed frequent peanut consumption during pregnancy {OR, 2.9(95% CI, 1.7,4.9)} to be associated with peanut IgE ≥5 kUA/L. Chung Laboratory analysis After curing and roasting, mature peanuts exhibited approximately 20% higher levels of advanced glycation end adducts and higher IgE binding vs immature peanuts. Yadzir Laboratory analysis Extracts from raw shrimp bound higher IgE than extracts from boiled shrimp, but the purified boiled tropomysoin (the main shrimp allergen) demonstrates higher IgE binding vs raw shrimp. Samson Laboratory Thermal processing can lead to the formation of new antigenic structures. Milner Cohort Early vitamin D use (within the first 6 months of life) was associated with a higher risk for food allergies in the exclusively formula-fed population [OR,1.63(95% CI,1.21,2.20)]. Vitamin use at 3 years of age was associated with increased risk for food allergies but not asthma in both breastfed [OR,1.62(95% CI,1.19,2.21) ]and exclusively formula-fed infants [OR, 1.39(95% CI,1.03,1.88)]. |

| | | States, with the highest rates found in New England. [adjusted β for New England vs the rest of the US, 4.07 (95%CI, 2.77,5.36)] | |
|---|---|---|---|
| Mulins et | Ecologic study | Using multivariate analysis, EpiPen prescription rates were higher in southern | (61) |
| al | | latitudes (less sunlight) compared with northern regions [ $\beta$ , $-19.22$ ( 95% CI, | |
| | | -26.71 , -11.73)]. | |
| Mulins et | Ecologic study | Southern latitudes were associated with higher hypoallergenic formulae | (62) |
| al | | prescription rates [beta, -147.98( 95% CI,-281.83 , -14.14)]. | |

OR, odds ratio;RR, Relative Risk; CI,confidence interval ;CMA, Cow's Milk Allergy

## Appendix B. protocols.

# Initial Egg Challenge/Desensitization doses (12)\*:

| Dose (n:0) | Mg egg protein | Dosage form |
|------------|----------------|--------------------------------------|
| 1 | 0.1 | Excipient microcrystalline cellulose |
| 2 | 0.2 | |
| 3 | 0.4 | "<br>— — |
| 4 | 0.8 | "<br>—— |
| 5 | 1.5 | "<br>— — |
| 6 | 3 | -"- |
| 7 | 6 | "<br>— — |
| 8 | 12 | Dose of the powder |
| 9 | 25 | "<br>— — |
| 10 | 50 | "<br>— — |
| 11 | 75 | "<br>— — |
| 12 | 100 | "<br>—— |
| 13 | 125 | "<br>— — |
| 14 | 150 | "<br>—— |
| 15 | 200 | |
| 16 | 250 | "<br>— — |

| 17 | 300 |
|----|-----|

Increasing doses are given approximately every 30 minutes. If the subject does not tolerate a given dose and symptoms are mild, then that dose or the previously tolerated one is repeated, and the protocol proceeds as outlined. If the subject experiences significant symptoms, then the protocol is stopped, and the highest tolerated dose is used as the starting daily dose.

**Post – Escalation Egg challenge (Egg Protein):** 

| Number of dose | Egg protein mg at | <b>Cumulative dose</b> |
|----------------|-------------------|------------------------|
| | dose | |
| 1 | 1mg | 1 |
| 2 | 3mg | 4 |
| 3 | 10mg | 14 |
| 4 | 30mg | 44 |
| 5 | 100mg | 144 |
| 6 | 300mg | 443 |
| 7 | 600mg | 1043 |
| 8 | 1000mg | 2043 |
| 9 | 2000mg | 4043 |
| 10 | 2000mg | 6043 |

10 doses of powdered Meringue given every 10 to 20 minutes in increasing amounts up to a total of 10 g of powdered egg white (6.04 g of egg protein which is equivalent to 1 egg).

Scale for Grading Reaction Severity and management

| Score | Symptom | Action |
|---|---|---|
| Mild | Pruritus, | Observe |
| | Urticaria, | May give Antihistamine (e.g. |
| | Flushing, | Benadryl or Reactin as prescribed |
| | Rhinoconjunctivitis | Call Research Team |
| | | Research team will evaluate if dose |
| | | adjustment is needed and if next dose |
| | | will be given at home or in hospital. |
| Moderate | Angioedema, | Give epinephrine IM as per protocol |
| | Throat tightness, | Give Antihistamine (e.g. Benadryl or |
| | Gastrointestinal complaints (cramping, | Reactin as prescribed |
| | . pain,vomiting,diarrhea) | Seek urgent care (hospital emergency |
| | Respiratory symptoms (Cough, Mucous | room) |
| | production) | Call Research team |
| | | To give next adjusted dose in hospital |
| | | research unit (CIM) |
| Severe | Wheeze, Respiratory Distress | Give epinephrine IM as per protocol |
| | Hypoxia, | Give Antihistamine (e.g. Benadryl or |
| | Cyanosis, | Reactin as prescribed |
| | Hypotension | Call 911 |
| | Circulatory collapse (Shock) | Seek urgent care (transfer to hospital |
| | | emergency room) |
| | | Call Research team; if the symptoms |
| | | are not improving within 10 minutes |
| | | of the first dose, instructions will be |
| | | given from the team regarding use of |
| | | a second dose of epinephrine. |

Appendix C. Budget

Total budget estimate: 78,000CAD per year including:

| Estimate (CAD) | comment |
|----------------|---------|

| Yearly salary for an | 35,000 | |
|---------------------------------------|--------|--------------------|
| undergraduate student for expenses | | |
| related to training in Lab evaluation | | |
| mechanisms for auto-immune | | |
| urticaria detection | | |
| Study coordinator | 40,000 | Yearly salary with |
| | | benefits |
| Paediatric test center (70CAD | 3000 | |
| for each blood sample) | | |
| Staining with monoclonal Abs | 3000 | |
| Use of FACS | 3000 | |
| CBA | 3500 | |
| Culture materials and stimulating | 3500 | |
| material | | |
| Travel expenses for presentation | 5000 | |
| of results in scientific conferences | | |
| | 78,000 | yearly |

Appendix D Study Schema

